CLINICAL TRIAL: NCT04938583
Title: Phase 1b/2, Single Arm Clinical Trial to Evaluate the Safety and Activity of Oregovomab and Bevacizumab, Paclitaxel Carboplatin as a Combinatorial Strategy in Subjects With BRCA-wild Type Platinum Sensitive Recurrent Ovarian Cancer
Brief Title: Oregovomab in Combination With Bevacizumab Plus Chemo in BRCA Wild Type Platinum Sensitive Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CanariaBio Inc. (Industry)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Jung KH, MD, Professor, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG GY20-10
Record Dates: First submitted 2021-05-24; First posted 2021-06-24 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer by FIGO Stage; Ovarian Cancer Stage III; Ovarian Cancer Stage IV
Keywords: Oregovomab; CA 125; platinum-sensitive recurrent ovarian cancer; bevacizumab; paclitaxel; carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — oregovomab; Bevacizumab; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- oregovomab, bevacizumab, paclitaxel and carboplatin (Experimental): Combination of anti-angiogenesis and Chemo-immunotherapy
  Interventions: Biological: Oregovomab; Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Oregovomab — Oregovomab will be administered on day1 cycle 1, 3, 5, and 9. A minimum of 3 patients will be enrolled into each cohort (2 mg or 1 mg).
  2 mg (starting dose), dissolved in 2 mL of 0.9% Sodium Chloride Injection USP, then added to 50 mL of Sodium Chloride Injection USP infused over 20 ± 5 minutes
  Other Names: MAb-B43.13
Drug: Bevacizumab — 15mg/Kg Day 1 (every 21 days) until progression
  Other Names: Avastin
Drug: Paclitaxel — 175 mg/m^2, Day 1 x 6 cycles (every 21 days)
  Other Names: Taxol, Paxcel, Padexol
Drug: Carboplatin — AUC 5 IV Day 1 x 6 cycles (every 21 days)
  Other Names: Neoplatin

SUMMARY:
This is a single arm phase 1b/2 evaluation of the combination of oregovomab, and bevacizumab, paclitaxel carboplatin in adult subjects with CA125-associated, advanced recurrent epithelial ovarian, fallopian tube or peritoneal carcinoma (FIGO Stage III/IV) with BRCA-wild type, previously treated with 1 prior lines of therapy, and with platinum free intervals of >6 months since last platinum-based treatment.

DETAILED DESCRIPTION:
This study is an open-label, single arm, phase 1b/II, multicenter study.

In phase 1b part, the recommended phase 2 dose of oregovomab combined with bevacizumab, paclitaxel and carboplatin will be examined. Approximately 3 to 12 subjects("3+3" dose finding design) will be enrolled in phase 1b trial with starting dose of 2mg oregovmab.

In Phase II trial, response rate of combination with oregovomab and bevacizumab, paclitaxel will be examined. Based on Simon's two stage model, 8 patients will be enrolled in first stage, after review of efficacy (response rate) of study treatment, 30 additional subjects for second stage of phase 2 will be enrolled. Considering 10% of screening failure rate, overall 42 patients will be enrolled in phase 2 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females (19 years old and older) with CA125-associated recurrent epithelial adenocarcinoma of ovarian, fallopian tube or peritoneal origin.
2. Have one of the eligible histologic epithelial cell types: serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, carcinosarcoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.).
3. Patients must have had a complete or partial response to front-line platinum-based therapy (at least three cycles) and a treatment -free interval without clinical evidence of progressive disease at least 6 months.
4. No known deleterious or pathogenic germline or somatic BRreast CAncer gene (BRCA) mutation
5. Must have had an elevated serum CA125 > 2 times of UNL measured at the first diagnosis or screening within 28 days of start of study treatment.
6. Must have measurable disease, including identification of marker lesions, by radiographic or physical criteria suitable for evaluation according to RECIST v1.1 for documentation of disease response or progression.
7. Must have a ECOG Performance Status of 0, 1 or 2
8. Must have adequate organ function defined as:

   1. neutrophil count ≥1000 μL
   2. platelet count ≥100,000 μL
   3. Hemoglobin >9.0 g/dl
   4. Serum creatinine <1.5 times the upper normal limits (UNL) or creatinine clearance > 45 mL/min/1.73 m2
   5. bilirubin <1.5 times the UNL
   6. SGOT and SGPT < 2 times the UL
9. Must have voluntarily agreed to participate and have signed the informed consent, and are willing to complete all study procedures.

Exclusion Criteria:

1. Patients who have received more than one line of chemotherapy (maintenance is not considered a second line)
2. Have an active autoimmune disease (e.g., rheumatoid arthritis, SLE, ulcerative colitis, Crohn's Disease, MS, ankylosing spondylitis) requiring continuing immune suppressive therapy
3. Use of immunosuppressants within 28 days prior to the first administration of the current or clinical trial drug. However, intranasal, inhalation, and systemic administration of prednisone 10 mg/day or a physiological dose not exceeding the equivalent dose of corticosteroids are recognized as exceptions.
4. Known allergy to murine proteins or have had a documented anaphylactic reaction to any drug, or a known hypersensitivity to diphenhydramine or other antihistamines of similar chemical structure.
5. Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections (testing during the study is not mandatory).
6. Recognized immunodeficiency condition including human immunodeficiency virus (HIV) infection, cellular immunodeficiencies, hypogamma globulinemia or dysgammaglobulinemia; subjects who have acquired, hereditary, or congenital immunodeficiency's, including HIV infection
7. Patients with previous solid organ transplantation
8. Evidence of clinically significant cardiovascular conditions including uncontrolled hypertension, myocardial infarction within 1 year, uncontrolled or unstable angina, congestive heart failure (New York Heart Association Class III or IV), arrhythmia (Grade 2 or higher), chronic obstructive pulmonary disease, clinical significant proteinuria (>1g/24hr urine)
9. Patients with other invasive malignancies, with the exception of non-melanomatous skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates with this protocol.
10. Have ever previously received oregovomab or bevacizumab
11. Patients who received major surgical procedure within 28days
12. Pregnant or breast-feeding

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 1cycle (21days)
  Assessment of Dose Limiting toxicity (DLT) based on incidences and severity of adverse events will be measured according to CTCAE v5.0
Efficacy based on overall response rate (ORR) | Every 6 weeks (each cycle is 21 days)
  Overall response rate measured as the Percentage of Participants with a Complete Response (CR) or Partial Response (PR), as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECISTv1.1)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Date of randomization up until date of first documented disease progression or date of death from any cause, whichever comes first
  PFS, defined as date of first study treatment to the date of event defined as the first documented progression as per RECIST v1.1 or death due to any cause
Overall Survival (OS) | Date of randomization up until date of death from any cause
  OS, defined as date of first study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jung KH, MD, Principal Investigator — Asan Medical Hospital
Locations (6):
- South Korea (6):
  - Kyungpook National University Chilgok Hospital, Daegu
  - CHA Bundang Medical Center, Seongnam-si
  - Korea Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No